CLINICAL TRIAL: NCT01560247
Title: Percutaneous Recanalization in Ischemic Stroke Management in Europe Observational Registry
Acronym: PRIISM2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MindFrame, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: EU-PRIISM-02
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Revascularization; Mechanical thrombectomy; Neurothrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment Group: Subjects in whom a MindFrame Device was employed for restoration of flow and clot removal
  Interventions: Procedure: Mechanical thrombectomy

INTERVENTIONS:
Procedure: Mechanical thrombectomy — Mechanical thrombectomy using a MindFrame device
  Other Names: MindFrame; Capture; Flow

SUMMARY:
To determine the revascularization rate, clinical efficacy and safety of the CE-marked MindFrame System in ischemic stroke patients

DETAILED DESCRIPTION:
To determine the revascularization rate, clinical efficacy and safety in a "real-world setting" of the CE-marked MindFrame System in ischemic stroke patients with thrombotic neurovascular occlusions caused by an embolus deemed appropriate for endovascular treatment. Target vessels include the basilar, internal carotid and middle cerebral (M1 and M2 segments) arteries.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke for whom the physician has prescribed mechanical thrombectomy as appropriate therapy

Exclusion Criteria:

* Intracranial hemorrhage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The purpose of this registry is to compile data in a "real world setting". All subjects in whom there is an attempt to use the device will be included in the registry. All subjects must be recruited according to the Mindframe System "Instructions For Use".
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Procedural Efficacy | Immediate postprocedure
  The ability of the MindFrame System to restore blood flow by removing thrombus and establishing final Thrombolysis in Cerebral Infarction (TICI) 2b or 3 perfusion
Safety | 90 days postprocedure
  The rate of device-related serious adverse events
Clinical Efficacy | 90 days postprocedure
  The rate of modified Rankin Scale (mRS) score 0-2 at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soderman, MD, PhD, Principal Investigator — Karolinska Institutet